CLINICAL TRIAL: NCT02596633
Title: A Feasibility Randomized Control Trial (RCT) of Telephone-supported Acceptance and Commitment Therapy (ACT) for Low Mood in Multiple Sclerosis (MS)
Brief Title: A RCT of Telephone-supported ACT in MS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14094
Record Dates: First submitted 2015-10-16; First posted 2015-11-04 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants carry on with their usual care
- Intervention (Active Comparator): ACT self help book with telephone support calls; Telephone-support Acceptance and Commitment therapy (ACT)
  Interventions: Behavioral: Telephone-support Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Telephone-support Acceptance and Commitment Therapy (ACT) — Telephone-support Acceptance and Commitment Therapy (ACT): ACT self-help book and 8 telephone support calls
  Arms: Intervention

SUMMARY:
This study will investigate the feasibility of running a randomised controlled trial (RCT) of a psychotherapy called "Acceptance and Commitment Therapy (ACT)", delivered in a self-help format with additional telephone support from a therapist, for people with Multiple Sclerosis (MS) and low mood.

DETAILED DESCRIPTION:
A large proportion of people with Multiple Sclerosis (MS) suffer from emotional problems, therefore a large percentage of people with MS would be eligible to take part in a study offering a psychotherapeutic component to address these issues.

Acceptance and Commitment Therapy (ACT) has been found to be effective for mood problems, and been successfully used in self-help format, but no study has thus-far examined potential for use as an effective intervention in this (MS) population.

People will MS and low mood will be recruited from a neurology outpatient clinic. They will be randomized to either receive treatment as usual, or an ACT self-help book with 8 supportive telephone calls from a trainee clinical psychologist. Measures of anxiety, depression, quality of life and physical health will be administered at baseline, post-intervention and six month follow up. A sub sample of 10 participants will be interviewed to find out their view on taking part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS. Over 7 on the Hospital Anxiety and Depression Scale

Exclusion Criteria:

* Already receiving psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment, measured with telephone-interviews. | At post-intervention, which is the specific time point when participants report to the researchers that they have finished their self-help books and support calls, or exactly 12 weeks after randomisation for those in the treatment-as-usual arm
  A sub-sample of participants will be interviewed over the phone to assess their views on their recruitment into the trial.
Feasibility of randomisation, measured with telephone-interviews. | At post-intervention, which is the specific time point when participants report to the researchers that they have finished their self-help books and support calls, or exactly 12 weeks after randomisation for those in the treatment-as-usual arm
  A sub-sample of participants will be interviewed over the phone to assess their views on how they were randomised.
Feasibility of psychometric assessment, measured with telephone-interviews. | At post-intervention, which is the specific time point when participants report to the researchers that they have finished their self-help books and support calls, or exactly 12 weeks after randomisation for those in the treatment-as-usual arm
  A sub-sample of participants will be interviewed over the phone to assess their views on the battery of psychometric assessments.
Feasibility of the self-help book, measured with telephone-interviews. | At post-intervention, which is the specific time point when participants report to the researchers that they have finished their self-help books and support calls, or exactly 12 weeks after randomisation for those in the treatment-as-usual arm
  A sub-sample of participants will be interviewed over the phone to assess their views on the self-help book.
Feasibility of the telephone-support calls, measured with telephone-interviews. | At post-intervention, which is the specific time point when participants report to the researchers that they have finished their self-help books and support calls, or exactly 12 weeks after randomisation for those in the treatment-as-usual arm
  A sub-sample of participants will be interviewed over the phone to assess their views on the telephone support calls.

SECONDARY OUTCOMES:
Effectiveness in reducing anxiety, as measured using online psycho-metrics. | At post-intervention (12 weeks after randomisation) and 6 months after randomisation
  Effectiveness will be assessed using quantitative measures which will be completed by participants online.
Effectiveness in reducing depression, as measured using online psycho-metrics. | At post-intervention (12 weeks after randomisation) and 6 months after randomisation
  Effectiveness will be assessed using quantitative measures which will be completed by participants online.
Effectiveness in reducing physical health problems, as measured using online psycho-metrics. | At post-intervention (12 weeks after randomisation) and 6 months after randomisation
  Effectiveness will be assessed using quantitative measures which will be completed by participants online.
Effectiveness in increasing quality of life, as measured using online psycho-metrics. | At post-intervention (12 weeks after randomisation) and 6 months after randomisation
  Effectiveness will be assessed using quantitative measures which will be completed by participants online.

IPD SHARING:
Plan to Share IPD: No